CLINICAL TRIAL: NCT02800096
Title: Online Interventions for Problem Gamblers With and Without Co-occurring Mental Health Concerns: Randomized Controlled Trial
Brief Title: Online Interventions for Gamblers With and Without Co-occurring Mental Health Concerns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 004/2015
Record Dates: First submitted 2016-06-08; First posted 2016-06-15 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Gambling; Depression; Anxiety
MeSH Terms: conditions — Gambling; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gambling Internet intervention (Active Comparator): The gambling only Internet intervention (G-only) will consist of a new online version of self-change tools that have previously been translated successfully into an online form and shown to have a significant impact on gambling in three trials. A major focus of this intervention is to provide individuals with clear and concise behavioral and cognitive strategies for meeting the goal of reducing or quitting gambling.
  Interventions: Behavioral: Gambling Internet intervention
- Gambling Internet intervention + MoodGYM (Experimental): The G+MH intervention condition will consist of the G-only intervention and an online intervention for depression and anxiety. The mental health intervention chosen is MoodGYM, an extensively evaluated intervention found to be effective in a variety of different settings.
  Interventions: Behavioral: Gambling Internet intervention; Behavioral: MoodGYM

INTERVENTIONS:
Behavioral: Gambling Internet intervention — The gambling Internet intervention consists of a new online version of self-change tools that have previously been translated successfully into an online form and shown to have a significant impact on gambling in three trials. A major focus of this intervention is to provide individuals with clear and concise behavioral and cognitive strategies for meeting the goal of reducing or quitting gambling.
Behavioral: MoodGYM — Internet intervention for depression and anxiety - MoodGYM, an extensively evaluated intervention found to be effective in a variety of different settings.
  Arms: Gambling Internet intervention + MoodGYM

SUMMARY:
Comorbidity between problem gambling and mental health concerns such as anxiety and depression is common. Further, the treatment needs of people with co-occurring gambling and mental health concerns may be different from those of problem gamblers who do not have a co-occurring mental health concern. The present study is a two-arm, double blinded, parallel group randomized controlled trial (RCT) that will evaluate whether there is a benefit to providing access to mental health Internet interventions (G+MH intervention) in addition to an Internet intervention for problem gambling (G-only intervention) in participants with gambling problems who do or do not have co-occurring mental health concerns.

DETAILED DESCRIPTION:
People with gambling concerns will be recruited using targeted advertisements. Potential participants will be screened using an online survey to identify participants meeting criteria for problem gambling. As part of the baseline screening process, measures of current depression and anxiety will be assessed. Eligible participants agreeing to take part in the study will be randomized to one of two versions of an online intervention for gamblers - an intervention that just targets gambling issues (G-only) versus one that contains interventions for anxiety and depression in addition to an intervention for gamblers (G+MH). It is predicted that problem gamblers who do not have co-occurring mental health concerns will display no significant difference between intervention conditions at a six-month follow-up. However, for those with co-occurring mental health concerns, it is predicted that participants receiving access to G+MH website will display significantly reduced gambling outcomes at six-month follow-up as compared to those provided with G-only website.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* Score of 3 or greater on the Problem Gambling Severity Index of the Canadian Problem Gambling Index (PGSI- CPGI)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
The NORC DSM-IV Screen for Gambling Problems (NODS) past 3 month version indicating DSM-IV gambling severity. | 3 and 6 months
  Change in gambling severity (NODS) from baseline

SECONDARY OUTCOMES:
Number of days gambled per month | 3 and 6 months
  Change in mean days per month gambling from baseline

CONTACTS AND LOCATIONS:
Overall Officials: John A Cunningham, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Najavits LM, Ledgerwood DM, Afifi TO. A Randomized Controlled Trial for Gambling Disorder and PTSD: Seeking Safety and CBT. J Gambl Stud. 2023 Dec;39(4):1865-1884. doi: 10.1007/s10899-023-10224-z. Epub 2023 Jun 12. PMID 37306874
- [Derived] Cunningham JA, Hodgins DC, Mackenzie CS, Godinho A, Schell C, Kushnir V, Hendershot CS. Randomized controlled trial of an Internet intervention for problem gambling provided with or without access to an Internet intervention for co-occurring mental health distress. Internet Interv. 2019 Mar 6;17:100239. doi: 10.1016/j.invent.2019.100239. eCollection 2019 Sep. PMID 30906694
- [Derived] Cunningham JA, Hodgins DC, Bennett K, Bennett A, Talevski M, Mackenzie CS, Hendershot CS. Online interventions for problem gamblers with and without co-occurring mental health symptoms: Protocol for a randomized controlled trial. BMC Public Health. 2016 Jul 22;16:624. doi: 10.1186/s12889-016-3291-7. PMID 27449527
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.ca/en/research